CLINICAL TRIAL: NCT02320006
Title: Effect of Acupuncture on Incomplete Fallopian Tube Obstructive Infertility: Study Protocol for Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Liu (Other)
Responsible Party: Sponsor-Investigator, Li Liu, LiLiu, First Affiliated Hospital of Heilongjiang Chinese Medicine University
Organization: First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstHeilongjiang
Record Dates: First submitted 2014-12-14; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Female Infertility Due to Occlusion of Fallopian Tube
Keywords: hydrotubation; incomplete fallopian tube obstructive infertility; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- True acupuncture plus hydrotubation (Active Comparator): The treatment group will receive true acupuncture and hydrotubation,Hydrotubation (80,000 U gentamicin , 400U chymotrypsin , 5mg dexamethasone , 50ml 0.9% saline) will be performedwithin 3 7 days after the menstruation[12].We use a manometer to measure the pressure and record the number on a card, then calculate the gap of the first and last time,it continues 3 menstrual cycles. The points (points used for every participant of treatment group) include bilateral RN4、CV6、CV3、EX-CA1、ST36、SP6,All the needles will be keep in positions for 30 min.Acupuncture will be performed three times per week,for a total of 36 sessions (12 wk)
  Interventions: Other: acupuncture
- control acupuncture plus hydrotubation (Sham Comparator): The control group will receive control acupuncture and hydrotubation.Hydrotubation (80,000 U gentamicin , 400U chymotrypsin , 5mg dexamethasone , 50ml 0.9% saline) will be performed within 3 7 days after the menstruation[12].We use a manometer to measure the pressure and record the number on a card, then calculate the gap of the first and last time,it continues 3 menstrual cycles.Two needles will be inserted in each arm, one in each shoulder and one in each upper arm at nonacupuncture pointsAll the needles will be keep in positions for 30 min. Acupuncture will be performed three times per week,for a total of 36 sessions (12 wk).
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — For RN4、CV6 CV3 and EX-CA1, needles will be inserted vertically to the abdominal muscles. The acupuncturist can feel resistance from the tip of the needle when touching the muscles and continues to insert it to a depth of 2-3 mm and stops. For ST36 and SP6, needles will be inserted vertically to a depth of 25 mm. The needles will be manipulated with an even lifting and twisting method three times to achieve the sensation of deqi.

SUMMARY:
Acupuncture is one of the traditional Chinese practices widely used in China for more than 3000 years. In recent years, the use of acupuncture within infertility has gained popularity all over the world, but there is no research describing the use of acupuncture in infertility of incompletely obstructive fallopian tube. In this paper, we present a research design evaluating the effects of acupuncture on incomplete fallopian tube obstructive infertility. This is a randomized, control acupuncture and signal-blind trial. A total of 120 patients will be enrolled in this study and will be randomized into two groups. True acupuncture plus hydrotubation or control acupuncture plus hydrotubation will be performed for 12 weeks. The purpose of this paper is to evaluate the additional value of acupuncture on the tubal patency rate and pregnancy rate beyond Hydrotubation ,therefore to guide clinical.

ELIGIBILITY:
Inclusion Criteria:

* I.Patients between 22 and 42 years of age with infertility II.diagnosis of incomplete Fallopian tube obstruction based on one of the following conditions: a. Tubal patency test: Hydrotubation , Hysterosalpingography (HSG) or Hysterosonosalpingography (HSS) shows incomplete bilateral Fallopian tube obstruction b. Hysteroscopy: Hysteroscopic tubal cannulation hydrotubation proves bilateral tube incompletely patent. c. Laparoscopy: incomplete bilateral tubal obstruction can be displayed by the methylene blue solution through the tubes III.Other relative treatments are not carried out within two weeks IV.willing to cooperate with us V. mean infertility time is 1-5 years.

Exclusion Criteria:

* I.allergic constitution or be allergic to diatrizoate or a variety of drugs II.the infertility is not leaded by tubal obstruction ,such as Congenital Physiological defects or malformation, genetic factors, immune factors and endocrine factors III.diagnosed with uterine lesions by auxiliary examinations (endometriosis ,adenomyosis , hysteromyoma or cancer and so on ) and infertility caused by tubal tuberculosis IV. infertility factor in their male partner V.people with Serious primary diseases of cardiovascular, liver, kidney and hematopoietic systems ,patients with mental illness VI.unable to judge the therapeutic efficacy or incomplete information VII.complete bilateral tubal obstruction VIII.bilateral tubes patent IX.Not willing to give written consent to the study X. people who are pregnant XI.people with acute infection .

Ages: 22 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
tubal patency rate | 3 months

SECONDARY OUTCOMES:
pregnancy rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- LiLiu, Harbin, Heilongjiang, China